CLINICAL TRIAL: NCT01097759
Title: LigaSure Hemorrhoidectomy vs Stapled Hemorrhoidopexy: a Prospective Randomized Clinical Trial
Brief Title: LigaSure Hemorrhoidectomy Versus Stapled Hemorrhoidopexy
Status: Completed | Type: Observational
Sponsor: Kuwait Oil Company Ahmadi Hospital (Other)
Collaborators: Netherlands: Ministry of Health, Welfare and Sports (Other Government)
Responsible Party: Mohamed Moussa, Ahmadi Hospital
Other Study IDs: 58061302393
Record Dates: First submitted 2010-04-01; First posted 2010-04-02 (Estimated); Last update posted 2010-04-02 (Estimated); Status verified 2006-01

CONDITIONS: Prolapsed Hemorrhoids
Keywords: hemorrhoids; prolapsed; hemorrhoidectomy; Hemorrhoidopexy; LigaSure; Stapled
MeSH Terms: conditions — Hemorrhoids | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- LigaSure: LigaSure is a vascular sealing device that can seal the hemorrhoidal plexus during hemorrhoidectomy (surgery)
  Interventions: Procedure: Surgery
- Stapler: Circular stapler that removes excess loose tissue above the anus and interrupts the blood supply during hemorrhoidal surgery
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Surgery — Hemorrhoidectomy using the LigaSure sealing device or hemorrhoidopexy using the stapler

SUMMARY:
This study was designed to compare the outcome of LigaSure hemorrhoidectomy and stapled hemorrhoidopexy for prolapsed hemorrhoids.

DETAILED DESCRIPTION:
The study was designed as a single-blind, prospective, randomized controlled trial and was approved by the Ethics Committee of Ahmadi Hospital, Kuwait. Patients were randomly assigned to undergo either hemorrhoidectomy with the LigaSure device or stapled hemorrhoidopexy. Patients were blinded as to the type of procedure perform. Candidates for the study were consecutive patients with symptomatic grade III or IV hemorrhoids admitted to the Ahmadi Hospital (secondary care hospital), Kuwait, from January 2006 through July 2007.

ELIGIBILITY:
Inclusion Criteria:

* Adult (above 18 years)
* With prolapsed hemorrhoids (grades III or IV)

Exclusion Criteria:

* Complicated hemorrhoid
* Coexisting perianal disease
* Previous perianal surgery
* Unfit for general anesthesia
* Pregnancy
* History of bleeding tendency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 68 patients with symptomatic grade III or grade IV hemorrhoids entered the study.
Sampling Method: Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2006-01; Primary Completion 2007-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Assessment of postoperative pain | 12 months
  Postoperative pain was assessed using the visual analogue scale (VAS)

SECONDARY OUTCOMES:
Assessment of postoperative complications | 12 months
  Postoperative complications and their management were compared between both groups during the followup visits for 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud F Sakr, MD, PhD, Principal Investigator — Professor of Surgery, Faculty of Medicine, Alexandria University
Locations (1):
- Ahmadi Hospital, Al Ahmadi, Al Ahmadi, Kuwait